CLINICAL TRIAL: NCT03482076
Title: Prevelance of Iron Deficiency Anemia in Liver Cirrhosis in Childern
Brief Title: Iron Deficiency Anemia in Childern With Liver Cirrhosis
Acronym: IDA
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Bahaa Khaled Mohamed Mohamed, assistant lecturer, Assiut University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: DBK
Record Dates: First submitted 2018-03-23; First posted 2018-03-29 (Actual); Last update posted 2018-03-29 (Actual); Status verified 2018-03

CONDITIONS: Iron Deficiency, Anaemia in Children; Liver Cirrhosis
MeSH Terms: conditions — Iron Deficiencies; Liver Cirrhosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- transferrin receptor concentration (Other): Prevelance of iron deficiency in this patients
  Interventions: Diagnostic Test: transferrin receptor concentration

INTERVENTIONS:
Diagnostic Test: transferrin receptor concentration — Sandwich radio-imunoassay

SUMMARY:
Iron deficiency anemia is a common complication of liver cirrhosis in childern and may affects there life this study to improve the outcome of these patients

DETAILED DESCRIPTION:
Patients with cirrhosis are at risk of developing both IDA and anemia of chronic disease concomitantly, and there adverse effects can deteriorate general condition and affect of quality of life in these patients .Also because it is easier to correct IDA than anemia of chronic disease, so this study of the prevalence of IDA helping us in the diagnosis and treatment of IDA and can reduce the need for other diagnostic tests and improve the quality of life in patients with cirrhosis .

ELIGIBILITY:
Inclusion Criteria:

* all childern with liver cirrhosis in GIT and hepatology unit

Exclusion Criteria:

* Neonates less than one month
* childern with other liver diseases

Ages: 1 Month to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 50 (Estimated)
Dates: Start 2019-03-01 (Estimated); Primary Completion 2020-03-01 (Estimated); Study Completion 2020-06-01 (Estimated)

PRIMARY OUTCOMES:
Prevelance of IDA in liver cirrhosis | two years
  To evaluate results